CLINICAL TRIAL: NCT04964908
Title: CREEK is a Multicenter Retrospective Study to Understand the Clinical Characteristics, Treatment Pathway and Resource Utilization for Patients With Chronic Lymphocytic Leukemia in International Region.
Brief Title: Study to Understand Clinical Characteristics, Treatment Pathway in Chronic Lymphocytic Leukemia
Acronym: CREEK
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00031
Record Dates: First submitted 2021-07-08; First posted 2021-07-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Multicenter Retrospective Study to understand the clinical characteristics, treatment pathway and resource utilization for patients with chronic lymphocytic leukemia A retrospective, multi-centre, observational study to describe disease characteristics, treatment patterns, treatment-related outcomes, and resource utilization for Chronic Lymphocytic Leukemia (CLL) patients in multiple international regions

DETAILED DESCRIPTION:
CREEK is a retrospective, observational, registry-based study including patients with an incidental diagnosis of CLL and started treatment (1st line, 2nd line, or Subsequent lines of treatment) within the period between 01 June 2016 and 12 months before data collection as identified from the patient records (from participating hospitals across the GCC States and the International region countries) with at least 12 months of follow-up, after starting on treatment.

Moreover, the study will include a pilot cohort in the GCC as an exploratory objective to describe the clinical and patient characteristics for the treatment-naive CLL patient

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Chronic Lymphocytic Leukemia (CLL)
* Initiated CLL treatment (including 1st line, 2nd line, or Subsequent lines of treatment) within the period between 01 June 2016, and 12 months before data collection

  - For GCC pilot cohort patients: treatment-naive CLL patients diagnosed between 01 June 2016, and 12 months before data collection.
* Available medical records at the participating site reflecting at least 12 months of follow-up after starting on treatment (except in the case of the participant death within one year following treatment initiation).
* Provision of informed consent by the patient or next of kin/legal representative (for deceased patients at study entry, unless a waiver was granted), according to local regulations.
* Adult male or female ≥18 years old at the time of diagnosis or according to the age of majority as defined by local regulations).

Exclusion Criteria:

* Failure to meet one or more of the inclusion criteria.
* Any diagnosis of B-cell malignancies other than CLL.
* Current or prior use of "acalabrutinib" treatment.
* Currently/previously receiving treatment in an interventional clinical trial at the time of entry into this study for indications CLL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: with chronic lymphocytic leukemia (CLL) subjects diagnosed
Sampling Method: Probability Sample
Enrollment: 1088 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
To describe the clinical characteristics for with chronic lymphocytic leukemia (CLL) patients | 5 year
  To describe the clinical characteristics for with chronic lymphocytic leukemia (CLL) patients, recording the patient characteristic:
  - Demographics: (Age, gender, race, nationality, Performance status, Tobacco use, Family history of malignancies)
Calculation of Epidemiological Measure(s) of Interest | 5 years
  Calculation of Epidemiological Measure(s) of Interest e.g., descriptive statistics, hazard ratios, incidence rates, test/retest reliability)
To describe the clinical characteristics for with chronic lymphocytic leukemia (CLL) patients | 5 Years
  To describe the clinical characteristics for with chronic lymphocytic leukemia (CLL) patients, recording the patient characteristic:
  * Laboratory Status:
    * CBC: Hemoglobin, Total leucocytic count, neutrophils, lymphocytes, and platelets
    * Renal functions: serum creatinine, Urea, eGFR
    * Hepatic function: ALT and AST
  * Concomitant medications:
    * Antagonists of vitamin K
    * Oral Anticoagulants: rivaroxaban, apixaban, dabigatran
    * Proton pump inhibitors (PPIs)
    * H2 Antagonists
    * Antacids
    * Others
To describe the clinical characteristics for with chronic lymphocytic leukemia (CLL) patients | 5 Years
  To describe the clinical characteristics for with chronic lymphocytic leukemia (CLL) patients, recording the patient characteristic:
  * Comorbidities.
  * Risk stratification
To describe disease Characteristics | 5 Years
  To describe Staging of disease, Prognosis, Cytogenetics abnormalities and Immunogenetic analysis
  * Date of diagnosis
  * Staging of disease
To describe disease Characteristics | 5 Years
  To describe Staging of disease, Prognosis, Cytogenetics abnormalities and Immunogenetic analysis
  * Prognosis made by fluorescence in situ hybridization (FISH)
  * Immunogenetic analysis

SECONDARY OUTCOMES:
Recording the treatment patterns | 5 years
  Percentage of patients who received immediate therapy and median time of observation, Number of prior lines of treatment received.
Calculation of Epidemiological Measure(s) of Interest | 5 Years
  * First Treatment received:
  * Number of prior lines of treatment received
Subsequent lines of therapies | 5 Years
  Type of regimen (CIT or targeted therapies) and specific regimens or drugs
  * Number of cycles
  * Duration of treatment
  * Pattern of response at the end of the treatment

OTHER OUTCOMES:
Recording the treatment-related outcomes | 5 years
  Assessment of best response followed the IWCLL 2018 guidelines based on clinical description and biochemistry,

CONTACTS AND LOCATIONS:
Locations (41):
- Research Site, Buenos Aires, Argentina
- Brazil (3):
  - Research Site, Campinas
  - Research Site, Jaú
  - Research Site, São Paulo
- Research Site, Providencia, Chile
- Colombia (3):
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Medellín
- Research Site, San José, Costa Rica
- Research Site, Santo Domingo. D.N., Dominican Republic, Dominican Republic
- Egypt (3):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, Luxor
- India (9):
  - Research Site, Manipal, India
  - Research Site, Ahmedabad
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Haryāna
  - Research Site, Hyderabad
  - Research Site, Kashmīr
  - Research Site, Kolkata
  - Research Site, Mumbai
- Research Site, Kuwait City, Kuwait
- Malaysia (3):
  - Research Site, Kuala Selangor, Malaysia
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
- Mexico (2):
  - Research Site, Mexico City
  - Research Site, Monterrey
- Research Site, Panama City, Panama
- Saudi Arabia (2):
  - Research Site, Jeddah
  - Research Site, Riyadh
- Research Site, Singapore, Singapore
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Turkey (Türkiye) (6):
  - Research Site, Adana/Saricam, Turkey
  - Research Site, Izmir/ Bornova, Turkey
  - Research Site, Izmir/Balcova, Turkey
  - Research Site, Samsun/Atakum, Turkey
  - Research Site, Ankara/Altindag
  - Research Site, Ankara/Yenimahalle
- Research Site, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Url Preview for AstraZeneca Clinical Trials Website AstraZeneca Clinical Trials Website This web site provides clinical trial data, results and other information regarding clinical trials
  astrazenecagrouptrials.pharmacm.com
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Abdelmoaty M, Alshehri H, Alamoudi S, Buyukasik Y, Abdelfattah R, Alorabi M, Kamal A, Aboutaleb A, Alhejazi A. Chronic lymphocytic leukaemia in the Middle East: a subgroup analysis from the CREEK study on treatment patterns and outcomes. Expert Rev Anticancer Ther. 2025 Nov 11:1-12. doi: 10.1080/14737140.2025.2582649. Online ahead of print. PMID 41175395
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220R00031&attachmentIdentifier=f21390c7-0f86-4cf2-a143-ace5d944d7f8&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=